CLINICAL TRIAL: NCT05202340
Title: A Survey to Investigate Possible Factors That Will Affect the Choice of Androgen Deprivation Therapy in Prostate Cancer Patients
Brief Title: Factors Affecting Androgen Deprivation Therapy Choice in Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2021.492
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer: Patients diagnosed with prostate cancer
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of this study is to investigate possible factors that will affect the choice of androgen deprivation therapy in prostate cancer patients. This is a cross-sectional study performed in Prince of Wales Hospital in Hong Kong. One hundred patients will be recruited for this study.

DETAILED DESCRIPTION:
The incidence of prostate cancer in Hong Kong almost tripled between 1996 and 2010, with the highest increased incidence rate in total forms of malignancy. The incidence of prostate cancer in Hong Kong increased up to 28.9 per 100,000 men in 2017 (Age-standardized rate) (Hong Kong Cancer Registry 2017) and ranked third in all men cancers in Hong Kong. Certain environmental elements have had an effect on the increased rate of prostate cancer, including the transition to Western dietary habits and an aging population because of the rise in average life expectancy. In addition to environmental causes, the medical development of laboratory diagnoses and wide prostate-specific antigen usage in Hong Kong have also contributed to the increase in diagnosis of prostate cancer in recent years. Certainly, the efforts from different health bodies in public education about the condition have helped to raise public awareness about the condition, which also increase the pick-up of early disease in Hong Kong.

Androgen deprivation treatment (ADT) has become the standard treatment for metastatic prostate cancer in the past decades. Androgen deprivation can be achieved by three main modalities, namely bilateral orchidectomy, gonadotropin-releasing hormone (GnRH) agonist and GnRH antagonist. Apart from injectable ADT, oral GnRH antagonist has been approved recently. ADT can be different in terms of mechanism of action, route of drug administration (injection vs oral), site of injection and frequency of drug administration. Each different formulation may contribute to patient's choice on their drug usage [1-3]. However, information regarding the preference of choice and factors affecting the choice of ADT formulation were not available in the literature. Therefore, in this study, possible factors that will affect patient's choice of ADT, reason and preference on their ADT choice will be investigated.

The objective of this study is to investigate possible factors that will affect patient's choice of ADT therapy. This is a cross-sectional study performed in Prince of Wales Hospital in Hong Kong. One hundred patients will be recruited for this study.

After obtaining informed consent, trained research staffs will assist the subjects to perform this cross-sectional survey. Information related to patients' background (including, but not limited to: age, educational level, work-status, living situation), disease background (stage of disease), concomitant drug usage & administrative frequency, preference on drug usage (ADT vs injection; frequency of drug administration), history of ADT usage, reason and preference on their ADT choice, will be collected from the survey.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer only happens in male patients
* Patients who are currently receiving at least one dose of LHRH agonist or antagonist, as androgen deprivation therapy
* Patients who are willing to consent and participate in this study

Exclusion Criteria:

* Patients who received bilateral orchidectomy as androgen deprivation therapy
* Patients who, in the opinion of investigators, are not able to comprehend about the study questions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer only happens in male patients
Study Population: Patients diagnosed with prostate cancer in Prince of Wales Hospital will be identified in specialist clinics and then enrolled to the study,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Possible factors that will affect patient's choice of ADT therapy | 1 year
  Possible factors that will affect patient's choice of ADT therapy

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Psarou A, Cooper H, Wilding JPH. Patients' Perspectives of Oral and Injectable Type 2 Diabetes Medicines, Their Body Weight and Medicine-Taking Behavior in the UK: A Systematic Review and Meta-Ethnography. Diabetes Ther. 2018 Oct;9(5):1791-1810. doi: 10.1007/s13300-018-0490-5. Epub 2018 Aug 17. PMID 30120753
- [Background] Blackwood C, Sanga P, Nuamah I, Keenan A, Singh A, Mathews M, Gopal S. Patients' Preference for Long-Acting Injectable versus Oral Antipsychotics in Schizophrenia: Results from the Patient-Reported Medication Preference Questionnaire. Patient Prefer Adherence. 2020 Jul 2;14:1093-1102. doi: 10.2147/PPA.S251812. eCollection 2020. PMID 32753849
- [Background] Kane JM, Leucht S, Carpenter D, Docherty JP; Expert Consensus Panel for Optimizing Pharmacologic Treatment of Psychotic Disorders. The expert consensus guideline series. Optimizing pharmacologic treatment of psychotic disorders. Introduction: methods, commentary, and summary. J Clin Psychiatry. 2003;64 Suppl 12:5-19. PMID 14640142